CLINICAL TRIAL: NCT00322361
Title: A Study in Healthy Neonates of Safety, Tolerability, and Immunogenicity of Recombinant Hepatitis B Vaccine Manufactured Using a Modified Process
Brief Title: Modified Process Hepatitis B Vaccine in Healthy Neonates (V232-056)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V232-056; 2006_007
Record Dates: First submitted 2006-05-02; First posted 2006-05-05 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B; Hepatocellular Carcinoma
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Modified Process Hepatitis B Vaccine
  Interventions: Biological: Comparator: Modified process Hepatitis B Vaccine
- 2 (Active Comparator): Recombivax HB™
  Interventions: Biological: Comparator: RECOMBIVAX HB™

INTERVENTIONS:
Biological: Comparator: RECOMBIVAX HB™ — RECOMBIVAX HB™ 3 x 5-mcg regimen administered via intramuscular injection.
  Arms: 2
Biological: Comparator: Modified process Hepatitis B Vaccine — Modified Process Hepatitis B 3 x 5-mcg regimen administered via intramuscular injection.
  Arms: 1

SUMMARY:
Hepatitis B Vaccine [Recombinant] is a well-established vaccine which has been used extensively, worldwide since its initial licensure in 1986. Hepatitis B vaccines: [1] induce protection against the morbidity and mortality of acute hepatitis B virus infection, [2] reduce the incidence of chronic infection in vaccinated populations, and [3] thereby, reduce the incidence of hepatocellular carcinoma. The purpose of the trial is to assess if the new manufacturing process of the Hepatitis B Vaccine [Recombinant] vaccine shows the same level of hepatitis B antibody response or better as the currently licensed Hepatitis B Vaccine [Recombinant] vaccine. This study will also confirm that the new process vaccine is as well tolerated as the current vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female full-term (37-42 weeks gestation) neonates (birth to 10 days of age)
* Born to mothers with documented negative test for HBsAg within 9 months prior to delivery

Exclusion Criteria:

* Infant born to mother with no prenatal care
* Known or suspected impairment of immunologic function
* Prior vaccination with any hepatitis B vaccine for infant or mother(within 6 months prior to the birth of infant.)
* Recent(<72 hours) history of febrile illness >/= 99.5 degrees F (>/= 37.5 degrees C) axillary or >/= 100.5 degrees F (>/= 38.1 degrees C) rectal
* Any prior administration of hepatitis B immune globulin (HBIG), serum immune globulin, or any other blood-derived product, or the receipt by the mother of either immunoglobulin or HBIG within 6 months prior to birth of the infant
* Receipt of investigational vaccines by mother or infant within 3 months prior to first injection with study vaccine or if scheduled to be given to the infant during the study
* Known or suspected hypersensitivity to any component of study vaccine (e.g., aluminum, yeast)
* Any infant who cannot be adequately followed for study visits during the course of the clinical study
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 566 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer to hepatitis B surface antigen at Month 7 | 4 weeks Post Dose 3

SECONDARY OUTCOMES:
Safety and tolerability including use of Vaccination Report Card | Follow-up 14 days Post Vaccination 1, 2, & 3 (Via Vaccination Report Card)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Minervini G, McCarson BJ, Reisinger KS, Martin JC, Stek JE, Atkins BM, Nadig KB, Liska V, Schodel FP, Bhuyan PK. Safety and immunogenicity of a modified process hepatitis B vaccine in healthy neonates. Vaccine. 2012 Feb 14;30(8):1476-80. doi: 10.1016/j.vaccine.2011.12.095. Epub 2012 Jan 5. PMID 22227229
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html